CLINICAL TRIAL: NCT05330559
Title: Fluorescence, Light-microscopy, Ultrasound Integrated / Intraoperative Diagnosis to MAXimise Resection
Acronym: FLUID-MAX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: FLUID-MAX
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Patients With Radiological, Clinical and Anamnestic Picture Compatible With a New Diagnosis of Glioblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fluid MAX group — to evaluate and compare with the histopathological analysis the various margin-assessment systems, including ultrasound, florescence, brightfield vision, new optical filters and microscope image post-processing systems, for the treatment of High Grade Gliomas (HGGs)

SUMMARY:
The present study aims to evaluate and compare with the histopathological analysis the various margin-assessment systems, including ultrasound, florescence, brightfield vision, new optical filters and microscope image post-processing systems, for the treatment of High Grade Gliomas (HGGs)

DETAILED DESCRIPTION:
Extent of Resection represents the cornerstone of surgery in terms of improving the prognosis of the patient with High Grade Gliomas, but total removal of neoplastic tissue is prevented by the amount of infiltration that is undetectable either by traditional preoperative MRI techniques or by the naked eye during surgery. Several techniques are currently used to define margins in the surgical setting, but the literature available on them to date is mostly focused on the assessment of postoperative GTR (Gross Total Resection), which tends to underestimate neoplastic tissue infiltration.

The evaluation of the efficacy of these techniques in detecting tumour infiltration by comparing them with the histopathology response on intraoperative biopsies taken after the debulking phase of the neoplasm could overcome this sensitivity limitation.

The study therefore intends to develop an algorithm that allows to discern between tumour infiltration and healthy parenchyma by means of different margin-assessment techniques in order to maximise the extent of resection in patients with HGGs.

ELIGIBILITY:
Inclusion Criteria:

Patients with radiological, clinical and anamnestic picture compatible with a new diagnosis of Glioblastoma for whom there is an indication for cytoreductive surgery at the Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta.

Exclusion Criteria:

* Patients aged less than 18 years at the time of radiological diagnosis
* Patients who have received radiation therapy in the same area as the neoplasm of interest
* Patients contraindicated to 5-ALA administration
* Patients whose neoplasm is in close proximity to functionally eloquent areas (Primary Motor, Broca's, Wernicke's areas)
* Patients who have not given their consent to take part in the research

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by HGGs
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-08 (Estimated); Primary Completion 2023-04-08 (Estimated); Study Completion 2024-04-08 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | year 2
  Evaluation of Sensitivity and Specificity of individual techniques (bright field observation, 5-ALA FGS and ioUS) in detecting tumor infiltration quantified by histopathological examination.

SECONDARY OUTCOMES:
Secondary Outcome | year 2
  Conduct a feasibility study on the use of the above techniques in sequence described;

OTHER OUTCOMES:
third Outcome | year 2
  compare the performance of the new Glow400 fluorescence technique with the traditional FL400 in identifying tumor infiltration with respect to the examination histopathology
fourth Outcome | year 2
  identify histological and / or genetic characteristics capable of influencing the performance of margin assessment techniques

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro - Perin, MD - PhD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaichana KL, Jusue-Torres I, Navarro-Ramirez R, Raza SM, Pascual-Gallego M, Ibrahim A, Hernandez-Hermann M, Gomez L, Ye X, Weingart JD, Olivi A, Blakeley J, Gallia GL, Lim M, Brem H, Quinones-Hinojosa A. Establishing percent resection and residual volume thresholds affecting survival and recurrence for patients with newly diagnosed intracranial glioblastoma. Neuro Oncol. 2014 Jan;16(1):113-22. doi: 10.1093/neuonc/not137. Epub 2013 Nov 26. PMID 24285550
- [Background] Pino MA, Imperato A, Musca I, Maugeri R, Giammalva GR, Costantino G, Graziano F, Meli F, Francaviglia N, Iacopino DG, Villa A. New Hope in Brain Glioma Surgery: The Role of Intraoperative Ultrasound. A Review. Brain Sci. 2018 Nov 19;8(11):202. doi: 10.3390/brainsci8110202. PMID 30463249
- [Background] Mahboob S, McPhillips R, Qiu Z, Jiang Y, Meggs C, Schiavone G, Button T, Desmulliez M, Demore C, Cochran S, Eljamel S. Intraoperative Ultrasound-Guided Resection of Gliomas: A Meta-Analysis and Review of the Literature. World Neurosurg. 2016 Aug;92:255-263. doi: 10.1016/j.wneu.2016.05.007. Epub 2016 May 10. PMID 27178235
- [Background] Stepp H, Stummer W. 5-ALA in the management of malignant glioma. Lasers Surg Med. 2018 Jul;50(5):399-419. doi: 10.1002/lsm.22933. Epub 2018 May 8. PMID 29737540
- [Background] Kiesel B, Mischkulnig M, Woehrer A, Martinez-Moreno M, Millesi M, Mallouhi A, Czech T, Preusser M, Hainfellner JA, Wolfsberger S, Knosp E, Widhalm G. Systematic histopathological analysis of different 5-aminolevulinic acid-induced fluorescence levels in newly diagnosed glioblastomas. J Neurosurg. 2018 Aug;129(2):341-353. doi: 10.3171/2017.4.JNS162991. Epub 2017 Oct 27. PMID 29076783
- [Background] Del Bene M, Perin A, Casali C, Legnani F, Saladino A, Mattei L, Vetrano IG, Saini M, DiMeco F, Prada F. Advanced Ultrasound Imaging in Glioma Surgery: Beyond Gray-Scale B-mode. Front Oncol. 2018 Dec 3;8:576. doi: 10.3389/fonc.2018.00576. eCollection 2018. PMID 30560090
- [Result] D'Amico RS, Englander ZK, Canoll P, Bruce JN. Extent of Resection in Glioma-A Review of the Cutting Edge. World Neurosurg. 2017 Jul;103:538-549. doi: 10.1016/j.wneu.2017.04.041. Epub 2017 Apr 17. PMID 28427971
- [Result] Hervey-Jumper SL, Berger MS. Maximizing safe resection of low- and high-grade glioma. J Neurooncol. 2016 Nov;130(2):269-282. doi: 10.1007/s11060-016-2110-4. Epub 2016 May 12. PMID 27174197